CLINICAL TRIAL: NCT02978924
Title: Trans-spinal Direct Current Stimulation in Primary Orthostatic Tremor
Acronym: STOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: C16-26; 2016-A01202-49 (Registry Identifier: IDRCB)
Record Dates: First submitted 2016-11-22; First posted 2016-12-01 (Estimated); Last update posted 2025-09-02 (Actual); Status verified 2021-08

CONDITIONS: Primary Orthostatic Tremor
Keywords: spinal cord; tsDCS; 3D motion capture; EMG
MeSH Terms: conditions — Primary orthostatic tremor

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cathodal tsDCS (Active Comparator): 20 min of active treatment
  Interventions: Device: tsDCS
- Sham tsDCS (Sham Comparator): 20 min of sham treatment
  Interventions: Device: tsDCS

INTERVENTIONS:
Device: tsDCS — 20 min of treatment applied at the thoracic level (active electrode) with reference placed on the right shoulder

SUMMARY:
To explore the effect of cathodal tsDCS vs sham tsDCS in primary orthostatic tremor. The investigators hypothesize that cathodal tsDCS but not sham tsDCS would be able to restore both motor and sensory pathways of the spinal cord leading to functional improvements.

DETAILED DESCRIPTION:
Regain of function and improvement of motor skills is a major challenge in motor disorders in which spinal cord functions play a key role. The growing development of non-invasive brain stimulations in the past decade led to significant progress in the understanding of neuronal abnormalities in patients with movement disorders that opens up new vistas for experimental treatments. However, these treatments are currently limited due to their high cost and lack of possibility to use in outpatients. Recently, trans-spinal direct current stimulation (tsDCS) has emerged as a novel tool to modulate non-invasively spinal cord excitability. This may be an excellent alternative to epidural stimulation, the sole technique available up to now to alter spinal functions in an invasive fashion. The overall goal of this study is to assess the potential of tsDCS to restore spinal cord functions in patients with primary orthostatic tremor (POT), a disorder with little or no current therapeutic resources and high disability for patients.

Using a crossover, randomized, double-blinded approach, cathodal (2mA, 20 min) or sham tsDCS (with the active electrodes over the thoracic level and the reference electrode on the right shoulder) will be delivered to 15 patients with POT. The maximal time in upright position determined by a force platform, the cortical excitability assessed by transcranial magnetic stimulation (input / output curve of the tibialis anterior muscle and short-latency afferent inhibition) and EMG activities of lower extremity muscles will be measured before (PRE), immediately and 30 minutes after current offset (POST0 and POST30 respectively). Cathodal and sham tsDCS will be delivered in two different sessions with a washout period of at least 7 days. The investigators anticipate that cathodal tsDCS but not sham tsDCS will be able to modulate both sensory and motor functions in POT and will, in turn, lead to functional improvement.

ELIGIBILITY:
Inclusion Criteria:

* Patients with POT diagnosed since at least 1 year
* Normal neurological examination with the exception of POT
* Patients with or without treatment for TOP, or with treatment not sufficiently effective
* Affiliated with the French social security scheme, universal medical coverages (CMU), or an equivalent scheme
* Signed informed consent

Exclusion Criteria:

* Psychiatric or neurological conditions (with the exception of POT)
* Presence of potential tsDCS risk factors including an electrically, magnetically or mechanically activated implant (including cardiac pacemaker, epidural stimulation electrodes, etc.), an intravascular clip or any other electrically sensitive support system, damaged skin at the stimulation sites (i.e., skin with ingrown hairs, acne, razor nicks, wounds that have not healed, recent scar tissue, broken skin, etc.)
* Presence of TMS risk factor including cardiac pacemaker, history of epilepsy, traumatic brain injury with loss of consciousness, intracerebral clips, cochlear or ocular implants
* Pregnancy in women (as determined by a urine pregnancy test in pre-menopausal women), or lactating women or women planning pregnancy during the course of the study
* Patients enrolled in another biomedical research at the time of the study
* Participant who does not wish to be informed of any clinically relevant abnormalities (as determined by the investigators) identified during the course of the study
* Patient under guardianship or curatorship, or under judicial supervision

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-01-17 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11-28 (Actual)

PRIMARY OUTCOMES:
Change in maximal time in the upright position without support | Before (PRE) and immediately after current offset (POST0)
  Force plateform

SECONDARY OUTCOMES:
Quantitative assessment of tremor (EMG) | Before (PRE), immediately after (POST0) and 30min (POST30) current offset
Cortical excitability assessed by Transcranial Magnetic Stimulation | Before (PRE), immediately after (POST0) and 30min (POST30) current offset

CONTACTS AND LOCATIONS:
Overall Officials: Marie Vidailhet, MD, Principal Investigator — marie.vidailhet@psl.aphp.fr
Locations (1):
- Centre investigation clinique, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lamy JC, Varriale P, Apartis E, Mehdi S, Blancher-Meinadier A, Kosutzka Z, Degos B, Frismand S, Simonetta-Moreau M, Meunier S, Roze E, Vidailhet M. Trans-Spinal Direct Current Stimulation for Managing Primary Orthostatic Tremor. Mov Disord. 2021 Aug;36(8):1835-1842. doi: 10.1002/mds.28581. Epub 2021 Mar 27. PMID 33772851